CLINICAL TRIAL: NCT03139799
Title: Long-term Tablet-computer Based Casual Puzzle Video Game Intervention in Healthy Older and Cognitively Impaired Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2016-01281
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Mild Cognitive Impairment; Acquired Brain Injury; Cognitive Impairment; Healthy
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This study uses a 16-week, assessor blinded, randomized crossover design with two phases of treatment and three waves of measurement. Participants are randomly allocated to either the experimental (group T) or control intervention (group C). Group T will first receive the experimental and then the control intervention (T-C) while group C is given the opposite order of intervention (C-T). In phase I both groups take a baseline measurement (pre-test), then group T is given the casual puzzle game task (experimental intervention) while group C is performing the newspaper reading task (control intervention). After phase I (8 weeks) both groups are post-tested (mid-test). In phase II, groups are switched and the control group C is given the experimental intervention (casual puzzle game task) while the experimental intervention group T now serves as control. After phase II (16 weeks) both groups are post-tested again.
Who Masked: Outcomes Assessor
Masking Description: This study will include outcome assessor blinding as recommended in a publication on methodological quality criteria for cognitive rehabilitation research and computer game training in older adults (Bleakley et al., 2015; Cicerone, Azulay, & Trott, 2009).
  This will ensure that the person conducting the assessment of outcome measures will be unaware of the participant's treatment condition. For this purpose, a central randomization procedure will be used where a designated staff member not involved in the study will conduct and securely maintain the randomization, contact and allocate participants and use central methods (e.g. phone or secure computer) after the patient is enrolled. This way the treatment assignments are not revealed to the assessors when conducting the outcome assessments. The assessors will also be excluded from any activity pertaining to the intervention activities (e.g. instructing participants, distributing the tablet-computers).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puzzle Video Game Intervention (Experimental): Group T will first receive the experimental and then the control intervention (T-C) In phase I both groups take a baseline measurement (pre-test), then group T is given the casual puzzle game task (experimental intervention). After phase I (8 weeks) both groups are post-tested (mid-test). In phase II, groups are switched and the the experimental intervention group T now serves as control. After phase II (16 weeks) both groups are post-tested again.
  Interventions: Behavioral: Experimental - Puzzle Video Game Intervention; Behavioral: Control - Tablet Newspaper Reading Intervention
- Tablet Newspaper Reading Intervention (Active Comparator): Group C will first receive the the control intervention and then experimental and (C-T). In phase I both groups take a baseline measurement (pre-test), then group C is performing the newspaper reading task (control intervention). After phase I (8 weeks) both groups are post-tested (mid-test). In phase II, groups are switched and the control group C is given the experimental intervention (casual puzzle game task). After phase II (16 weeks) both groups are post-tested again.
  Interventions: Behavioral: Experimental - Puzzle Video Game Intervention; Behavioral: Control - Tablet Newspaper Reading Intervention

INTERVENTIONS:
Behavioral: Experimental - Puzzle Video Game Intervention — The psychological intervention consists of two custom-made versions of popular commercial casual puzzle video games (Flow Free, Big Duck Games LCC; Bejeweled, PopCap Games). The puzzle games are delivered on tablet-computers computer (12.9-inch tablet computer iPad Pro, Apple Inc., Cupertino, CA, USA).
Behavioral: Control - Tablet Newspaper Reading Intervention — The control intervention uses a newspaper/ magazine reading task that will be delivered to participants using the same device (iPad Pro) as in the experimental intervention. The newspaper/ magazine reading task will be running on the built-in Apple Newsstand application. Participants will be offered subscriptions for two newspapers and/or magazines that they are instructed to read following the same regime as in the experimental condition.

SUMMARY:
This study aims at investigating the effects of tablet-based puzzle video games on cognitive function and emotional well-being. This study extends preliminary findings of studies looking at short-term benefits of playing puzzle video games to a long-term intervention in healthy older adults and patients suffering from cognitive impairment due to mild cognitive impairment or acquired brain injury. To this end, the investigators compare two interventions: A tablet-based puzzle video games experimental intervention and a control intervention tablet newspaper-reading control intervention. This study uses a 16-week, assessor blinded, randomized crossover design with two phases of treatment and three waves of measurement. Participants are randomly allocated to either the experimental or control intervention for 8 weeks, then interventions are crossed over. Both groups receive both interventions in opposite order. At three time points (pre-, mid- and post-test) higher cognitive function and emotional well-being are tested using standardised neuropsychological tests and questionnaires.

DETAILED DESCRIPTION:
The focus of the current project is to examine the cognitive and emotional benefits of a casual puzzle video game (CPVG) intervention in healthy older adults (HOA), patients suffering from mild cognitive impairment (MCI) and acquired brain injury (ABI). Although there have only been a small number of studies specifically using CPVG interventions, recent studies were able to demonstrate the validity of CPVG in improving attentional and executive function and speed of processing (Oei & Patterson, 2013; Stroud & Whitbourne, 2015; Styron, 2015) in healthy older adults as well as their potential in reducing depressive symptoms, physical stress and anxiety (Russoniello, O'Brien, & Parks, 2009). These findings match general findings from video game training studies reporting improved processing speed, attentional, executive and visuospatial skills (Jak et al., 2013). In addition a recent large-scale study showed that regular engagement in Sudoku and similar puzzles represents a cognitively enriching leisure activity prevents and delays age-related cognitive decline (Ferreira, Owen, Mohan, Corbett, & Ballard, 2015). Since depressive disorders affect between 10% and 20% older adults and even more in persons suffering from MCI and dementia, and that mood disorders affect about 31% (anxiety disorders up to 40%) patients after suffering a stroke, these populations could potentially draw both cognitive and emotional benefits from CPVG intervention (Arba et al., 2016; Barua, Ghosh, Kar, & Basilio, 2011; Robinson, 2003).

The main objective of this study is to investigate long-term training benefits of a CPVG intervention on cognitive and emotional functioning in healthy older adults and patients with cognitive impairment.

The primary objective of this study is to examine whether a long-term CPVG intervention significantly improves attentional function (visual search) and leads to in-game learning effects in healthy older participants and cognitively impaired patients (MCI, ABI). The secondary objectives include: a) improvements on further cognitive outcome measures proposed to be engaged by the CPVG (attention, processing speed, working memory and spatial reasoning) and b) the efficacy of the CPVG intervention in reducing symptoms of depression, anxiety and stress and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal visual acuity
* Informed consent as documented by signature
* Healthy older adults:
* Aged 65 years and older
* Absence of cognitive impairment as assessed with a Montreal Cognitive Assessment (MoCA) of above 26.
* Mild cognitive impairment:
* Aged 65 years and older
* Objective cognitive impairment as assessed with a Montreal Cognitive Assessment (MoCA) smaller than 26 (MoCA < 26).
* Acquired brain injury:
* Diagnosis of acquired brain damage and cognitive impairment (e.g. attentional and executive deficits) as diagnosed through neuropsychological assessment combined with a MoCA score of 26 and smaller

Exclusion Criteria:

* Insufficient coordinative, motor and perceptual ability to handle a tablet- computer.
* Healthy older adults: History of neurological or psychiatric deficits
* Acquired brain injury: History of any other psychiatric deficits
* Mild cognitive impairment: History of any other neurological or psychiatric deficits

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure - Attention: Visual Search | Pre-test (Baseline, week 0)
  Visual Scanning subtest from the computerized Test of Attentional Performance (TAP) test battery
Primary outcome measure - Attention: Visual Search | Mid-test (Change from Baseline at week 4)
  Visual Scanning subtest from the computerized Test of Attentional Performance (TAP) test battery
Primary outcome measure - Attention: Visual Search | Post-test (Change from Baseline at week 8)
  Visual Scanning subtest from the computerized Test of Attentional Performance (TAP) test battery

SECONDARY OUTCOMES:
Additional attentional outcomes | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Trail Making Test (TMT) Part A for selective attention and Part B for divided attention
Processing speed | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Pattern Comparison Test (PCT) for spatial perception speed as well as TMT-A and -B for visual search speed.
Working memory | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV) subtests Digit Span (forward, backward and complex) for verbal working memory, Spatial Span (forward and backward) for visuospatial working memory and Spatial Addition for complex visuospatial memory based on the n-back paradigm.
Spatial reasoning | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Maze Task from the Neuropsychological Assessment Battery (NAB) for planning, organization, reasoning and problem solving.
Emotion and well-being 1 | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Profile of Mood States (POMS) that measures six mood subscales
Emotion and well-being 2 | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  State Trait Anxiety Inventory (STAI) that measures anxiety as an emotional state and personality trait
Emotion and well-being 3 | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  World Health Organization's WHOQOL-BREF quality of life assessment
Self-efficacy | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Assessed with the General Self-Efficacy Scale
Intervention compliance | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  The data saved each time the participants engage in a session of the casual puzzle game intervention will serve as a measure of gameplay frequency and intervention compliance.
Game experience | Pre-test (Baseline, week 0), Mid-test (Change from Baseline at week 4) and Post-test (Change from Baseline at week 8)
  Measured with the Perception of Training Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Prabitha Urwyler, PD. Dr., Principal Investigator — University of Bern
Locations (1):
- ARTORG Center for Biomedical Engineering Research, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oei AC, Patterson MD. Enhancing cognition with video games: a multiple game training study. PLoS One. 2013;8(3):e58546. doi: 10.1371/journal.pone.0058546. Epub 2013 Mar 13. PMID 23516504
- [Background] Stroud MJ, Whitbourne SK. Casual Video Games as Training Tools for Attentional Processes in Everyday Life. Cyberpsychol Behav Soc Netw. 2015 Nov;18(11):654-60. doi: 10.1089/cyber.2015.0316. Epub 2015 Oct 8. PMID 26448498
- [Background] Russoniello CV, O'Brien K, Parks JM. EEG, HRV and Psychological Correlates while Playing Bejeweled II: A Randomized Controlled Study. Stud Health Technol Inform. 2009;144:189-92. PMID 19592761
- [Background] Jak AJ, Seelye AM, Jurick SM. Crosswords to computers: a critical review of popular approaches to cognitive enhancement. Neuropsychol Rev. 2013 Mar;23(1):13-26. doi: 10.1007/s11065-013-9226-5. Epub 2013 Feb 20. PMID 23423553
- [Background] Ferreira N, Owen A, Mohan A, Corbett A, Ballard C. Associations between cognitively stimulating leisure activities, cognitive function and age-related cognitive decline. Int J Geriatr Psychiatry. 2015 Apr;30(4):422-30. doi: 10.1002/gps.4155. Epub 2014 Jul 3. PMID 24989949
- [Background] Arba F, Ali M, Quinn TJ, Hankey GJ, Lees KR, Inzitari D; VISTA Collaboration. Lacunar Infarcts, Depression, and Anxiety Symptoms One Year after Stroke. J Stroke Cerebrovasc Dis. 2016 Apr;25(4):831-4. doi: 10.1016/j.jstrokecerebrovasdis.2015.12.018. Epub 2016 Jan 14. PMID 26778600
- [Background] Barua A, Ghosh MK, Kar N, Basilio MA. Prevalence of depressive disorders in the elderly. Ann Saudi Med. 2011 Nov-Dec;31(6):620-4. doi: 10.4103/0256-4947.87100. PMID 22048509
- [Background] Bleakley CM, Charles D, Porter-Armstrong A, McNeill MD, McDonough SM, McCormack B. Gaming for health: a systematic review of the physical and cognitive effects of interactive computer games in older adults. J Appl Gerontol. 2015 Apr;34(3):NP166-89. doi: 10.1177/0733464812470747. Epub 2013 Jan 17. PMID 24652863
- [Background] Cicerone KD, Azulay J, Trott C. Methodological quality of research on cognitive rehabilitation after traumatic brain injury. Arch Phys Med Rehabil. 2009 Nov;90(11 Suppl):S52-9. doi: 10.1016/j.apmr.2009.05.019. PMID 19892075